CLINICAL TRIAL: NCT00024622
Title: Positron Emission Tomography (PET) Scanning in Dopamine Disorders: Parkinson's Disease and Schizophrenia
Brief Title: PET Scanning in Parkinson s Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010232; 01-M-0232
Record Dates: First submitted 2001-09-23; First posted 2001-09-24 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-11-18

CONDITIONS: Schizophrenia; Parkinson's Disease
Keywords: Neurological Disorder; Regional Cerebral Blood Flow; Dopamine; Schizophrenia; Parkinson's Disease; Natural History; PD; Parkinson; Healthy Control; HV; Normal Control
MeSH Terms: conditions — Schizophrenia; Parkinson Disease; Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy volunteers: Healthy volunteers.
  Interventions: Drug: O-15 Water
- Patients - Parkinsons: Patients with Parkinsons
  Interventions: Drug: 18F-Fluoro-L-dopa; Drug: O-15 Water
- Patients - schizophrenia spectrum disorders: Patients - schizophrenia spectrum disorders
  Interventions: Drug: 18F-Fluoro-L-dopa; Drug: O-15 Water

INTERVENTIONS:
Drug: 18F-Fluoro-L-dopa
  Groups: Patients - Parkinsons; Patients - schizophrenia spectrum disorders
Drug: O-15 Water

SUMMARY:
This is an in vivo positron emission tomography (PET) study of regional cerebral dopamine and blood flow in normal volunteers, persons with Parkinson s disease (both familial and sporadic), and those with schizophrenia spectrum disorders. The latter also sign consent for NIH approved protocol 89-M-0160, "Inpatient Evaluation of Neuropsychiatric Patients," PI: Daniel Eisenberg, M.D. Using PET with 6-[F-18] Fluoro-L-dopa (FDOPA) and (15)0-H2O in a single scan session, both presynaptic dopaminergic function and regional cerebral blood flow (rCBF) are assessed. The kinetic rate constant (Ki) for presynaptic dopaminergic uptake in striatum and other regions is calculated. We compare Ki across subject groups and relate the findings to rCBF. Findings are also related to allelic variation in genes of interest, for determination of which participants sign separate consent for NIH approved protocol 95-M-0150 Neurobiological Investigation of Patients with Schizophrenia Spectrum Disorders and Their Siblings, PI: Karen F. Berman, MD. We also draw comparisons between subjects with inherited vs. sporadic Parkinson s disease to determine whether the PET phenotype is the same in both groups, and we compare system-level, circuit-based pathophysiology across PD and schizophrenia groups. Each subject is further screened with an MRI to rule out structural abnormalities and also to further delineate areas of interest in the PET scans....

DETAILED DESCRIPTION:
This is an in vivo positron emission tomography (PET) study of regional cerebral dopamine and blood flow in normal volunteers, persons with Parkinson s disease (both familial and sporadic), and those with schizophrenia spectrum disorders. The latter also sign consent for NIH approved protocol 89-M-0160, "Inpatient Evaluation of Neuropsychiatric Patients," PI: Daniel Eisenberg, M.D. Using PET with 6-[F-18] Fluoro-L-dopa (FDOPA) and (15)0-H2O in a single scan session, both presynaptic dopaminergic function and regional cerebral blood flow (rCBF) are assessed. The kinetic rate constant (Ki) for presynaptic dopaminergic uptake in striatum and other regions is calculated. We compare Ki across subject groups and relate the findings to rCBF. Findings are also related to allelic variation in genes of interest, for determination of which participants sign separate consent for NIH approved protocol 95-M-0150 Neurobiological Investigation of Patients with Schizophrenia Spectrum Disorders and Their Siblings, PI: Karen F. Berman, MD. We also draw comparisons between subjects with inherited vs. sporadic Parkinson s disease to determine whether the PET phenotype is the same in both groups, and we compare system-level, circuit-based pathophysiology across PD and schizophrenia groups. Each subject is further screened with an MRI to rule out structural abnormalities and also to further delineate areas of interest in the PET scans.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age between 18 and 90 years
* Ability to give informed consent
* Ability to read and write
* Ability to give adequate medical and neuropsychiatric history.

PARKINSONS DISEASE:

* Individuals over the age of 18 from families in which an autosomal dominant form of Parkinson's disease is suspected based on pedigree analysis.
* Each subject will have a medical history and brief neurological examination.
* The diagnosis in probands must be supported by accepted clinical criteria: tremor, bradykinesia, and responsiveness to L-DOPA.
* Equivocally affected individuals will also be included in order to aid in their phenotypic classification as will at risk individuals who show no neurological signs.
* Individuals with sporadic Parkinson's disease will also be scanned. These will be over the age of 50 years and will have no known family history of Parkinson's disease or any other movement disorder.
* PD patients will have an admission physical exam and medical history as well as laboratory tests deemed necessary on the basis of history and physical exam.

SCHIZOPHRENIA:

- Members of this patient group will have a diagnosis of schizophrenia or schizophrenia spectrum disorder as determined by the SCID and will be currently enrolled in NIH approved protocol 89-M-0160 (Inpatient Evaluation of Neuropsychiatric Patients) under which they will have received admission work-up.

HEALTHY VOLUNTEERS:

* A large cohort of healthy volunteers will also have a PET scan.
* Volunteers will be age, gender and handedness-matched to patients for statistical purposes.
* Volunteers, who are enrolled as healthy controls under protocol 95-M-0150 "Neurobiological Investigation of Patients with Schizophrenia Spectrum Disorders and their Siblings" will receive admission workup through that protocol.

EXCLUSION CRITERIA:

* Will include medical illness that would affect cerebral blood flow or dopamine
* Current pregnancy
* Current breast feeding
* Possible exposure to radiation exceeding RSC guidelines
* History of any (excepting nicotinerelated) DSM5-defined moderate to severe substance use disorder (or DSM-IV-defined substance dependence).
* Cumulative lifetime history of any (excepting nicotine-related) DSM5-defined mild substance use disorder (or any DSM-IV-defined substance abuse),either in excess of 5 years total or not in remission for at least 6 months,
* Inability to stay caffeine- and nicotine-free for 4 hours
* Current suicidality or assaultiveness
* History of movement disorder
* History of head injury requiring hospitalization
* History of coma
* Inability to meet general safety criteria for MRI study (as determined by standardized Nuclear Medicine Research (NMR) Center screening)
* Previously demonstrated inability or unwillingness to comply with a study protocol.

PARKINSONS DISEASE:

- Individuals not capable of understanding the consent will be excluded.

HEALTHY VOLUNTEERS:

- Healthy volunteers will be unable to participate if they have been treated with psychotropic medication within the three months prior to scanning, are undergoing current psychiatric treatment, have any history of major psychiatric or movement disorder, have a first degree relative with schizophrenia, or have a family history of PD.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is an in vivo positron emission tomography (PET) study of regional cerebral dopamine and blood flow in normal volunteers, persons with Parkinson's disease (both familial and sporadic), and those with schizophrenia spectrum disorders.
Sampling Method: Probability Sample
Enrollment: 502 (Actual)
Dates: Start 2002-03-15 (Actual)

PRIMARY OUTCOMES:
To explore with positron emission tomography (PET) the pathophysiology and cerebral consequences of dopaminergic dysregulation. | Ongoing
  To explore with positron emission tomography (PET) the pathophysiology and cerebral consequences of dopaminergic dysregulation.

CONTACTS AND LOCATIONS:
Overall Officials: Karen F Berman, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Ianni AM, Eisenberg DP, Boorman ED, Constantino SM, Hegarty CE, Gregory MD, Masdeu JC, Kohn PD, Behrens TE, Berman KF. PET-measured human dopamine synthesis capacity and receptor availability predict trading rewards and time-costs during foraging. Nat Commun. 2023 Sep 30;14(1):6122. doi: 10.1038/s41467-023-41897-0. PMID 37777515
- [Derived] Eisenberg DP, Kohn PD, Hegarty CE, Smith NR, Grogans SE, Czarapata JB, Gregory MD, Apud JA, Berman KF. Clinical correlation but no elevation of striatal dopamine synthesis capacity in two independent cohorts of medication-free individuals with schizophrenia. Mol Psychiatry. 2022 Feb;27(2):1241-1247. doi: 10.1038/s41380-021-01337-1. Epub 2021 Nov 17. PMID 34789848
- [Derived] Eisenberg DP, Kohn PD, Hegarty CE, Ianni AM, Kolachana B, Gregory MD, Masdeu JC, Berman KF. Common Variation in the DOPA Decarboxylase (DDC) Gene and Human Striatal DDC Activity In Vivo. Neuropsychopharmacology. 2016 Aug;41(9):2303-8. doi: 10.1038/npp.2016.31. Epub 2016 Feb 29. PMID 26924680
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2001-M-0232.html